CLINICAL TRIAL: NCT06974669
Title: The Value of Using Mini-oral Pulse Steroid Therapy Along With Non Cultured Epidermal Cell Suspension in Stable Resistant Vitiligo: An Interventional Prospective Controlled Trial.
Brief Title: The Value of Using Mini-oral Pulse Steroid Therapy Along With Non Cultured Epidermal Cell Suspension (NCES) in Stable Resistant Vitiligo
Acronym: NCES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mogawer, Lecturer of Dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VS-OMP
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Vitiligo
Keywords: vitiligo; surgery; mini-oral pulse steroid therapy; resistant
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitiligo surgery with added mini-oral pulse steroid therapy in the peri-surgical period (Active Comparator): this group will receive oral mini-pulse steroids (low-dose dexamethasone: 5mg/week on 2 successive days per week) for 2 weeks prior to NCES and for 4 weeks afterwards
  Interventions: Drug: oral steroid-dexamethasone; Procedure: non cultured epidermal suspension
- Vitiligo surgery without mini-oral pulse steroid therapy (Active Comparator): this group will undergo None cultured epidermal suspension (NCES) without oral mini-pulse steroids.
  Interventions: Procedure: non cultured epidermal suspension

INTERVENTIONS:
Drug: oral steroid-dexamethasone — this study is the first according to the best of our knowledge assessing the value of adding mini oral pulse steroid therapy to non cultured epidermal suspension in treatment of stable acral and difficult to treat vitiligo
  Arms: Vitiligo surgery with added mini-oral pulse steroid therapy in the peri-surgical period
Procedure: non cultured epidermal suspension — this is the best surgical technique for surgical treatment of vitiligo that would be done for both arms

SUMMARY:
Assessing the additive value of mini-oral pulse steroid therapy in surgical treatment of acral and difficult to treat sites of vitiligo

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo (NSV) with acral or resistant lesions over the elbows and knees, that has not responded to conventional treatment
* Stability for ≥ 1 year
* Age ≥18 years
* Lack of topical treatment for at least 1 month prior to surgery and systemic treatment for at least 3 months prior to surgery.

Exclusion Criteria:

* Non acral NSV responsive to conventional treatment modalities
* Active vitiligo; new lesions, expansion of old lesions, confetti like lesions, ill-defined edges or koebnerization in < 1 year
* Age < 18 years.
* Pregnant females.
* Patients with hypertension, diabetes or tuberculosis
* Topical treatment in the past month and systemic treatment in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
comparing percent change in pigmentation in both arms | 3 months
  • Comparing percent change of pigmentation as per VESTA score after 3 months of treatment with NCES with and without mini oral pulse steroids.
comparing percent change in surface area in both arms | 3 months
  • Comparing percent change in the surface area of the depigmented patch following NCES using point counting technique.

SECONDARY OUTCOMES:
comparing physician global assessment in both arms | 3 months
  • Comparing physician global assessment after treatment with NCES with and without oral mini-pulse therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mogawer, MD, PhD, Principal Investigator — Dermatology Department, Cairo University Hopsitals
Locations (1):
- Dermatology Department, Cairo University Hospitals, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participants' data that underlie reported results will be shared upon request, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 3 months and for 12 months after completion of the study
Access Criteria: Controlled Access:
  Researchers who provide a methodologically sound proposal will be allowed to access data to achieve aims in the approved proposal